CLINICAL TRIAL: NCT07280286
Title: Incidence of Intrauterine Adhesions Following Myomectomies With the Use of an Intrauterine Anti-adhesion Gel
Brief Title: Incidence of Intrauterine Adhesions After Myomectomy With Intrauterine Anti-Adhesion Gel
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Brunella Zizolfi, PhD, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KE5DXJL9Z1F5
Record Dates: First submitted 2025-11-22; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Myoma;Uterus; Adhesion; Uterus, Internal
Keywords: intrauterine adhesions; myomectomy
MeSH Terms: conditions — Myofibroma; Tissue Adhesions; Gynatresia

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a prospective, randomized, non-profit trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Anti-adhesion gel group (Experimental): Women will receive the application of an anti-adhesion gel at the end of the myomectomy procedure.
  Interventions: Device: Women will receive the application of an anti-adhesion gel at the end of the myomectomy procedure
- Standard of care group (No Intervention): Women will not receive any anti-adhesion methods

INTERVENTIONS:
Device: Women will receive the application of an anti-adhesion gel at the end of the myomectomy procedure — The difference compared to other studies published in the past is that, in our trial, at the end of the robotic myomectomy-which will be performed using the same technique in both groups-an anti-adhesion gel will be applied in the intervention group to prevent the formation of intrauterine adhesions.
  Arms: Anti-adhesion gel group

SUMMARY:
This prospective randomized study aims to evaluate whether the application of an intrauterine anti-adhesion gel reduces the incidence of intrauterine adhesions (IUAs) following robotic-assisted laparoscopic myomectomy. Intrauterine adhesions may develop after endometrial trauma during surgery and can negatively affect menstrual function, fertility, and future pregnancy outcomes. Robotic myomectomy offers a minimally invasive approach, but postoperative adhesion formation remains a concern.

Sixty-two women undergoing myomectomy will be randomized to receive either intrauterine anti-adhesion gel (intervention group) or no adhesion-prevention method (control group). Adhesions will be assessed by ultrasound and hysteroscopy during follow-up. Secondary outcomes include reproductive results over a 24-month period, such as implantation rate, clinical pregnancy, miscarriage, live birth, pregnancy complications, and neonatal outcomes.

The study seeks to determine whether combining a minimally invasive surgical approach with an intrauterine gel provides additional protection against adhesion formation and improves fertility-related outcomes.

DETAILED DESCRIPTION:
Intrauterine adhesions (IUAs), or uterine synechiae, are fibrotic bands that develop when the endometrium is damaged and the normal healing process is disrupted. Surgical trauma-particularly involving the basal layer of the endometrium-is one of the main triggers for adhesion formation. Myomectomy is recognized as the gynecologic procedure most frequently associated with the development of adhesions, which may compromise uterine function, menstrual regularity, fertility, and obstetric outcomes. Although minimally invasive approaches such as conventional or robot-assisted laparoscopy have reduced postoperative morbidity, they cannot eliminate the risk of adhesion formation, especially when the uterine cavity is entered or extensive suturing is required.

Adhesion formation results from excessive fibrin deposition and insufficient fibrinolytic activity during tissue repair. When fibrin persists on the injured surfaces, fibroblast proliferation and neovascularization may lead to permanent fibrotic bridges between areas that should remain separated. This process is particularly relevant following myomectomy, where the endometrium may be inadvertently injured. Several studies have reported high rates of intrauterine adhesions after open myomectomy and, to a lesser extent, after minimally invasive procedures. Adhesions may occur even when the cavity is not breached, suggesting that the myometrial trauma itself can contribute to this pathological process.

Anti-adhesion gels have been proposed as an adjunctive strategy to prevent postoperative synechiae. These sterile, absorbable, highly viscous hydrophilic gels-typically composed of sodium carboxymethylcellulose (CMC), polyethylene oxide (PEO), and electrolytes-act as temporary mechanical barriers, physically separating traumatized surfaces during the healing period. Evidence from previous studies suggests that intrauterine gel application after hysteroscopic procedures may reduce adhesion formation and improve postoperative reproductive outcomes. However, few trials have evaluated the efficacy of these gels after laparoscopic or robotic myomectomy.

This study is a prospective, randomized, controlled, non-profit clinical trial designed to assess whether the application of an intrauterine anti-adhesion gel at the end of robotic-assisted laparoscopic myomectomy reduces the incidence of IUAs compared with no adhesion-prevention method. Sixty-two women undergoing myomectomy will be randomized 1:1 into an intervention group (with gel application) or a control group (without gel). All participants will undergo standardized preoperative assessment, including ultrasound and office hysteroscopy. Postoperative follow-up includes ultrasound at one month to evaluate pelvic adhesions and diagnostic hysteroscopy at two months to assess intrauterine adhesions. Reproductive outcomes will be monitored for up to 24 months through spontaneous or assisted conception attempts.

The primary endpoint is the incidence of intrauterine adhesions at follow-up hysteroscopy. Secondary endpoints include clinical pregnancy rate, implantation rate, miscarriage rate, live birth rate, pregnancy complications, mode of delivery, and neonatal outcomes.

The study aims to clarify whether combining a minimally invasive robotic approach with an intrauterine gel can synergistically reduce adhesion formation and improve fertility outcomes. Results may contribute to optimizing postoperative management in women undergoing myomectomy and refining strategies to preserve reproductive potential.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years;
* BMI 18-35;
* One or more fibroids diagnosed via ultrasound;
* First myomectomy or uterine surgery;
* Incomplete reproductive plans and/or infertility;
* Adequate immune, respiratory, liver, cardiac, bone marrow, and kidney function;
* Compliance and psychological ability to follow study procedures;
* Acceptance and signing of informed consent.

Exclusion Criteria:

* Age under 18 years;
* Age over 46 years;
* Pregnancy or breastfeeding;
* History of intrauterine adhesions;
* Diagnosis or suspicion of malignant gynecological pathologies and/or autoimmune diseases;
* Completed reproductive plans;
* Severe respiratory, bone marrow, liver, or kidney dysfunction preventing safe surgical access.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2026-04-06 (Estimated); Study Completion 2028-11-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy of intrauterine gel in reducing the formation of intrauterine adhesions | Up to two months after surgery
  The primary objective of the study is to evaluate the efficacy of intrauterine gel in reducing the formation of intrauterine adhesions following robotic-assisted laparoscopic myomectomy. Intrauterine adhesions will be assessed during follow-up ultrasound performed one month after surgery and by diagnostic hysteroscopy two months after surgery. Adhesions will be classified according to an internationally recognized scoring system. The severity, extent, and type of adhesions will be documented using the American Fertility Society (AFS) / American Society for Reproductive Medicine (ASRM) classification system, which categorizes IUAs as mild, moderate, or severe based on the extent of cavity involvement, type of adhesions, and menstrual pattern.

SECONDARY OUTCOMES:
Clinical Pregnancy Rate | Up to 24 months after surgery
  Presence of a gestational sac with fetal heartbeat detected on transvaginal ultrasound.
  Measurement: Confirmed by ultrasound between the 5th and 7th weeks of gestation and recorded in clinical data.
Live Birth Rate (LBR) | Up to 24 months post-surgery.
  Percentage of patients delivering a live-born infant after conception. Measurement: Collected from hospital records or via follow-up phone interviews
Miscarriage Rate | Up to 24 months after surgery
  Spontaneous pregnancy loss before 20 weeks of gestation. Measurement: Confirmed by ultrasound or clinical documentation in case of spontaneous abortion.
Pregnancy Complications | Up to 24 months after surgery
  Adverse events during pregnancy, such as gestational hypertension, preeclampsia, gestational diabetes, or preterm birth.
  Measurement: Collected from medical charts, obstetric reports, or standardized questionnaires.
Mode of delivery | Up to 24 months after surgery
  Type of delivery (spontaneous vaginal, assisted vaginal, cesarean section). Measurement: Recorded from birth certificates or hospital delivery records.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmes DR Jr. New devices versus conventional balloon technology in patients with coronary artery disease. J Interv Cardiol. 1992 Mar;5(1):47-9. doi: 10.1111/j.1540-8183.1992.tb00823.x. No abstract available. PMID 10150951
- [Background] Dargent D. [Indications for hysterectomy]. Contracept Fertil Sex. 1998 Jan;26(1):35. No abstract available. French. PMID 9532880
- [Background] Asgari Z, Hafizi L, Hosseini R, Javaheri A, Rastad H. Intrauterine synechiae after myomectomy; laparotomy versus laparoscopy: Non-randomized interventional trial. Iran J Reprod Med. 2015 Mar;13(3):161-8. PMID 26000007
- [Background] Lagana AS, Garzon S, Dababou S, Uccella S, Medvediev M, Pokrovenko D, Babunashvili EL, Buyanova SN, Schukina NA, Shcherbatykh Kaschchuk MG, Kosmas I, Licchelli M, Panese G, Tinelli A. Prevalence of Intrauterine Adhesions after Myomectomy: A Prospective Multicenter Observational Study. Gynecol Obstet Invest. 2022;87(1):62-69. doi: 10.1159/000522583. Epub 2022 Feb 15. PMID 35168241
- [Background] Capmas P, Pourcelot AG, Fernandez H. Are synechiae a complication of laparotomic myomectomy? Reprod Biomed Online. 2018 Apr;36(4):450-454. doi: 10.1016/j.rbmo.2018.01.010. Epub 2018 Feb 2. PMID 29454580
- [Background] Pellicano M, Guida M, Bramante S, Acunzo G, Di Spiezio Sardo A, Tommaselli GA, Nappi C. Reproductive outcome after autocrosslinked hyaluronic acid gel application in infertile patients who underwent laparoscopic myomectomy. Fertil Steril. 2005 Feb;83(2):498-500. doi: 10.1016/j.fertnstert.2004.09.019. PMID 15705404
- [Background] Acunzo G, Guida M, Pellicano M, Tommaselli GA, Di Spiezio Sardo A, Bifulco G, Cirillo D, Taylor A, Nappi C. Effectiveness of auto-cross-linked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic adhesiolysis: a prospective, randomized, controlled study. Hum Reprod. 2003 Sep;18(9):1918-21. doi: 10.1093/humrep/deg368. PMID 12923149
- [Background] Guida M, Acunzo G, Di Spiezio Sardo A, Bifulco G, Piccoli R, Pellicano M, Cerrota G, Cirillo D, Nappi C. Effectiveness of auto-crosslinked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic surgery: a prospective, randomized, controlled study. Hum Reprod. 2004 Jun;19(6):1461-4. doi: 10.1093/humrep/deh238. Epub 2004 Apr 22. PMID 15105384
- [Background] Pellicano M, Bramante S, Cirillo D, Palomba S, Bifulco G, Zullo F, Nappi C. Effectiveness of autocrosslinked hyaluronic acid gel after laparoscopic myomectomy in infertile patients: a prospective, randomized, controlled study. Fertil Steril. 2003 Aug;80(2):441-4. doi: 10.1016/s0015-0282(03)00597-1. PMID 12909511
- [Background] Sheng Y, Hong Z, Wang J, Mao B, Wu Z, Gou Y, Zhao J, Liu Q. Efficacy and safety of robot-assisted laparoscopic myomectomy versus laparoscopic myomectomy: a systematic evaluation and meta-analysis. World J Surg Oncol. 2023 Jul 28;21(1):230. doi: 10.1186/s12957-023-03104-8. PMID 37507735
- [Background] Di Saverio S, Coccolini F, Galati M, Smerieri N, Biffl WL, Ansaloni L, Tugnoli G, Velmahos GC, Sartelli M, Bendinelli C, Fraga GP, Kelly MD, Moore FA, Mandala V, Mandala S, Masetti M, Jovine E, Pinna AD, Peitzman AB, Leppaniemi A, Sugarbaker PH, Goor HV, Moore EE, Jeekel J, Catena F. Bologna guidelines for diagnosis and management of adhesive small bowel obstruction (ASBO): 2013 update of the evidence-based guidelines from the world society of emergency surgery ASBO working group. World J Emerg Surg. 2013 Oct 10;8(1):42. doi: 10.1186/1749-7922-8-42. PMID 24112637
- [Background] Moris D, Chakedis J, Rahnemai-Azar AA, Wilson A, Hennessy MM, Athanasiou A, Beal EW, Argyrou C, Felekouras E, Pawlik TM. Postoperative Abdominal Adhesions: Clinical Significance and Advances in Prevention and Management. J Gastrointest Surg. 2017 Oct;21(10):1713-1722. doi: 10.1007/s11605-017-3488-9. Epub 2017 Jul 6. PMID 28685387
- [Background] Beyene RT, Kavalukas SL, Barbul A. Intra-abdominal adhesions: Anatomy, physiology, pathophysiology, and treatment. Curr Probl Surg. 2015 Jul;52(7):271-319. doi: 10.1067/j.cpsurg.2015.05.001. Epub 2015 Jun 9. No abstract available. PMID 26258583
- [Background] Okabayashi K, Ashrafian H, Zacharakis E, Hasegawa H, Kitagawa Y, Athanasiou T, Darzi A. Adhesions after abdominal surgery: a systematic review of the incidence, distribution and severity. Surg Today. 2014 Mar;44(3):405-20. doi: 10.1007/s00595-013-0591-8. Epub 2013 May 9. PMID 23657643
- [Background] Tabibian N, Swehli E, Boyd A, Umbreen A, Tabibian JH. Abdominal adhesions: A practical review of an often overlooked entity. Ann Med Surg (Lond). 2017 Jan 31;15:9-13. doi: 10.1016/j.amsu.2017.01.021. eCollection 2017 Mar. PMID 28203370
- [Background] De Wilde RL, Bakkum EA, Brolmann H, Crowe A, Koninckx P, Korell M, Lundorff P, Pistofidis G, Tchartchian G, Trew G, Wattiez A, Wallwiener M. Consensus recommendations on adhesions (version 2014) for the ESGE Adhesions Research Working Group (European Society for Gynecological Endoscopy): an expert opinion. Arch Gynecol Obstet. 2014 Sep;290(3):581-2. doi: 10.1007/s00404-014-3312-7. Epub 2014 Jun 24. No abstract available. PMID 24958350
- [Background] Vrijland WW, Jeekel J, van Geldorp HJ, Swank DJ, Bonjer HJ. Abdominal adhesions: intestinal obstruction, pain, and infertility. Surg Endosc. 2003 Jul;17(7):1017-22. doi: 10.1007/s00464-002-9208-9. Epub 2003 Mar 14. PMID 12632122
- [Background] Diamond MP, Freeman ML. Clinical implications of postsurgical adhesions. Hum Reprod Update. 2001 Nov-Dec;7(6):567-76. doi: 10.1093/humupd/7.6.567. PMID 11727865
- [Background] Tulandi T, Murray C, Guralnick M. Adhesion formation and reproductive outcome after myomectomy and second-look laparoscopy. Obstet Gynecol. 1993 Aug;82(2):213-5. PMID 8336866

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT07280286/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT07280286/ICF_001.pdf